CLINICAL TRIAL: NCT01225263
Title: Combined Statin and Vitamin D Therapy for Prophylactic Treatment of Episodic Migraine
Brief Title: Statin/Vitamin D & Migraine Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rami Burstein (Other)
Responsible Party: Sponsor-Investigator, Rami Burstein, Professor, Beth Israel Deaconess Medical Center
Organization: Beth Israel Deaconess Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2010P000118
Record Dates: First submitted 2010-09-30; First posted 2010-10-20 (Estimated); Results first posted 2016-01-26 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2015-12

CONDITIONS: Migraine
Keywords: Migraine disorders; Headache; Simvastatin; Vitamin D
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — Simvastatin; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Simvastatin and vitamin D (Experimental): Participants in this arm will receive simvastatin + vitamin D.
  Interventions: Drug: Simvastatin; Dietary Supplement: Vitamin D
- Placebo "Sugar Pill" (Placebo Comparator): Participants in this arm will take placebo pills, which look like the simvastatin and vitamin D. A placebo pill has no active medication in it, and is like taking a "sugar pill".
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Simvastatin — simvastatin, 20 mg, twice daily for 6 months
  Arms: Simvastatin and vitamin D
Dietary Supplement: Vitamin D — Vitamin D3, 1000 IU, twice daily for 6 months
  Arms: Simvastatin and vitamin D
Other: Placebo — Two placebo pills, taken twice daily for 6 months
  Arms: Placebo "Sugar Pill"

SUMMARY:
The investigators are studying if taking simvastatin and vitamin D together will help prevent episodic migraines. Simvastatin is an FDA approved drug that is typically used to treat high cholesterol and reduce the risk of stroke and heart attack. Vitamin D is a vitamin found in certain foods like some types of fish, and in nutritional supplements. This study is 9 months long. Some people who participate will receive simvastatin and vitamin D, and some people will receive a placebo. A placebo is a "sugar pill" that looks like medication but does not have any active ingredients in it.

The investigators hypothesize that taking vitamin D and simvastatin daily may reduce the number of migraines people who have episodic migraine get.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Have had migraines for at least 3 years
* Have between 4 and 15 migraines a month
* Able to speak and read the English language

Exclusion Criteria:

* Women who are pregnant or nursing, or planning on becoming pregnant in the next 10 months
* Individuals who have a had a heart attack, stroke, peripheral artery disease, atherosclerotic aortic disease, carotid artery disease, or diabetes
* individuals at high risk for cardiovascular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2010-09; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Buettner, MD, MPH, Principal Investigator — Beth Israel Deaconess Medical Center; Rami Burstein, PhD, Study Director — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Buettner C, Nir RR, Bertisch SM, Bernstein C, Schain A, Mittleman MA, Burstein R. Simvastatin and vitamin D for migraine prevention: A randomized, controlled trial. Ann Neurol. 2015 Dec;78(6):970-81. doi: 10.1002/ana.24534. Epub 2015 Nov 13. PMID 26418341

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the greater Boston area. All study visits took place at Beth Israel Deaconess Medical Center (Boston, MA).
Pre-assignment Details: Of 89 participants enrolled, 32 were excluded prior to randomization: 8 not interested; 8 lost to follow up; 7 had <4 migraine days/mo; 4 had chronic daily headache; 2 daily opioid use; 1 chronic pain; 1 using a statin; 1 using a medication contraindicated with statin. The remaining 57 participants completed a 12-wk baseline and were randomized.
Groups:
- Simvastatin and Vitamin D: Participants in this arm took Simvastatin 20 mg twice daily for 6 months plus Vitamin D3 1000 IU twice daily for 6 months.
- Placebo "Sugar Pill": Participants in this arm took placebo pills, which looked like the Simvastatin and Vitamin D. Two placebo pills were taken twice daily for 6 months.
Period: Weeks 1 to 12
Arm/Group | Simvastatin and Vitamin D | Placebo "Sugar Pill"
Started | 28 | 29
Completed | 28 | 29
Not Completed | 0 | 0
Period: Weeks 13 to 24
Arm/Group | Simvastatin and Vitamin D | Placebo "Sugar Pill"
Started | 28 | 29
Completed | 24 | 28
Not Completed | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Simvastatin and Vitamin D: Participants in this arm received Simvastatin 20 mg twice daily and Vitamin D3 1000 IU twice daily for 6 months.
- Placebo: Participants in this arm received placebo pills, which looked like the Simvastatin pill and Vitamin D pill. Two placebo pills were taken twice daily for 6 months
- Total: Total of all reporting groups
Arm/Group | Simvastatin and Vitamin D | Placebo | Total
Number analyzed (Participants) | 28 | 29 | 57
Age, Customized [Median (Inter-Quartile Range); unit: years]
  Age | 40 [23 to 46] | 28 [21 to 34] | 33 [21 to 44]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 25 | 52
  Male | 1 | 4 | 5
Race/Ethnicity, Customized [Number; unit: participants]
  Non-Hispanic White | 24 | 21 | 45
  Other | 4 | 8 | 12
Recorded Migraine Days/Past 3m, Median (Interquartile Range) [Median (Inter-Quartile Range); unit: days] | 25.5 [14.5 to 34.0] | 18.0 [14.0 to 23.0] | 20 [14.0 to 28.0]

OUTCOME MEASURES:

1. Primary Outcome: Migraine Frequency: Change From Baseline 12-week Period to Weeks 1 to 12
Time Frame: Weeks 1 to 12
Measure: Median (Inter-Quartile Range); unit: days
Groups:
- Placebo: Participants in this arm received placebo pills, which looked like the simvastatin and Vitamin D pills, taken twice daily for 6 months
Arm/Group | Simvastatin and Vitamin D | Placebo
Number analyzed (Participants) | 28 | 29
days | -8.0 [-15.0 to -2.0] | 1.0 [-1.0 to 6.0]

2. Primary Outcome: Migraine Frequency: Change From Baseline 12-week Period to Weeks 13 to 24
Time Frame: Weeks 13 to 24
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Simvastatin and Vitamin D | Placebo
Number analyzed (Participants) | 28 | 29
days | -9.0 [-13.0 to -5.0] | 3.0 [-1.0 to 5.0]

ADVERSE EVENTS:
Arm/Group | Simvastatin and Vitamin D | Placebo
Serious Adverse Events (participants affected / at risk) | 0/28 | 1/29
Other Adverse Events (participants affected / at risk) | 5/28 | 10/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Simvastatin and Vitamin D (N=28) | Placebo (N=29)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — 1 participant in the placebo group had a creatine kinase (CK) level of 37,780 IU/L. On inquiry, the participant had been vigorously exercising while taking multiple stimulant-containing dietary supplements. The participant experienced full recovery.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Simvastatin and Vitamin D (N=28) | Placebo (N=29)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Joint pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Myalgia (without CK elevation) (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Skin rash or itch (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No